CLINICAL TRIAL: NCT02579824
Title: A Phase I Ascending Dose and Exploratory Expansion Study of DS-3032b, an Oral MDM2 Inhibitor, in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Ascending Dose and Exploratory Expansion Study of DS-3032b, an Oral MDM2 Inhibitor, in Subjects With Relapsed and/or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: stopped prematurely
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Daiichi Sankyo UK Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0101; NCI-2015-01873 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Myeloma
Keywords: Myeloma; Relapsed and/or Refractory; Multiple Myeloma; MM; DS-3032b
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS-3032b (Experimental): Dose Escalation Phase: DS-3032b administered once daily by mouth on Days 1 - 21 of a 28 day cycle. Starting dose level 90 mg/day.
  Dose Expansion Phase: Starting dose level maximum tolerated dose from Dose Escalation Phase.
  Interventions: Drug: DS-3032b

INTERVENTIONS:
Drug: DS-3032b — Escalation DS-3032b starting dose level 90 mg/day administered once daily by mouth on Days 1 - 21 of a 28 day cycle. For Dose Expansion maximum tolerated dose from Dose Escalation Phase.

SUMMARY:
This is a 2 part study: Part 1 (dose escalation) and Part 2 (dose expansion).

The goal of Part 1 of this clinical research study is to find the highest tolerable dose of DS-3032b that can be given to patients with multiple myeloma (MM) that is relapsed (has come back) and/or refractory (has not responded to treatment).

The goal of Part 2 of this clinical research study is to continue to study the safety of the highest tolerable dose found in Part 1 of the study.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 3 groups of up to 6 participants each will be enrolled in Part 1 of the study, and up to 10 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of DS-3032b you receive will depend on when you join this study. The first group of participants will receive the lowest dose level of DS-3032b. Each new group will receive a higher dose of DS-3032b than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of DS-3032b is found.

If you are enrolled in Part 2, you will receive DS-3032b at the highest dose that was tolerated in Part 1.

Study Drug Administration:

You will take DS-3032b capsules by mouth 1 time each day on Days 1-21 of each 28-day study cycle. On Days 1, 8, and 15 of Cycle 1, you will take your morning dose of study drug at the clinic.

You should take each dose of DS-3032b with at least 4 ounces of water about 2 hours before or 1 hour after a meal. If you miss or vomit a dose of study drug at home, you should not retake the missed or vomited dose. Wait and take the next scheduled dose.

You should bring any empty bottles and unused study drug to the clinic at each visit. You will be given a diary to record when you take your study drug each day.

Study Visits:

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 4 tablespoons) and urine will be collected for routine tests and to check the status of the disease.
* You will have an EKG.
* Blood (about 1 tablespoon) will be drawn for biomarker testing before your dose of study drug.

If you have had some of these tests performed recently, you may not need to have them repeated.

On Day 8 of Cycle 1:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* Blood (about 1 tablespoon) will be drawn for pharmacokinetic (PK) and biomarker testing before your dose of study drug. PK testing measures the amount of study drug in the body at different time points.

On Day 15 of Cycle 1:

* You will have a physical exam.
* Blood (about 2 tablespoons) and urine will be collected for routine tests.
* You will have an EKG.

On Day 1 of Cycle 2:

* You will have a physical exam.
* Blood (about 4 tablespoons) and urine will be collected for routine tests and to check the status of the disease.
* You will have a bone marrow biopsy/aspiration to check the status of the disease and for biomarker testing. You may have this procedure performed at anytime between Day 24 of Cycle 1 and Day 5 of Cycle 2.

On Days 8 and 15 of Cycle 2, blood (about 2 tablespoons) will be drawn for routine tests.

On Day 1 of Cycle 3:

* You will have a physical exam.
* Blood (about 4 tablespoons) and urine will be collected for routine tests and to check the status of the disease. If you can become pregnant, this routine blood or urine collection will include a pregnancy test.

On Day 1 of Cycles 4 and beyond:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn for routine tests and to check the status of the disease.
* If the doctor thinks it is needed, you will have a bone survey.
* If the doctor thinks it is needed, you will have a bone marrow biopsy and/or aspirate to check the status of the disease and for biomarker and cytogenetic testing.

Length of Study:

You may continue taking the study drug as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on this study will be over after you have completed follow-up.

End-of-Treatment Visit:

Within 30 days after your last dose of study drug:

* You will have a physical exam.
* Blood (about 4 tablespoons) and urine will be collected for routine tests and to check the status of the disease. If you can become pregnant, this routine collection will include a pregnancy test.

Follow-Up Visit:

About 30 days after your last dose of study drug, you will be contacted either by phone or during a clinic visit to find out what drugs you are taking and how you are doing. If you are called, it should take about 5 minutes.

This is an investigational study. DS-3032b is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 28 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have relapsed and/or refractory myeloma with measurable disease, as defined by at least one of the following: *Serum M-protein level >/=0.5 g/dL for Immunoglobulin G (IgG), Immunoglobulin A (IgA), or Immunoglobulin M (IgM) disease; * M-protein or total serum Immunoglobulin D (IgD) >/=0.5 g/dL for IgD disease; * Urinary Myeloma (M)-protein excretion of >/= 200 mg over a 24-hour period; * Involved free light chain level >/=10 mg/dL, along with an abnormal free light chain ratio.
2. Subjects must have had at least three lines of therapy for their disease, including a proteasome inhibitor and immunomodulatory drug (e.g., lenalidomide), with lines of therapy being separated by the presence of documented disease progression. Using this definition, treatment with induction therapy, followed by high dose chemotherapy and autologous stem cell transplantation, and finally by maintenance therapy, would constitute one line, provided that multiple myeloma did not meet criteria for progression at any time during this period.
3. Subjects must have disease that has relapsed and/or refractory after their most recent therapy, with progressive disease (PD) being defined as an increase of 25% from the lowest response value in any one or more of the following: *Serum M-protein (the absolute increase must be >/=0.5 g/dL) and/or; * Urine M-protein (the absolute increase must be >/=200 mg/24 hours) and/or; * Only in subjects without a measurable serum and urine M protein level: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase) must be >10 mg/dL; * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; * Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder.
4. Subjects with known polyneuropathy-organomegaly-endocrinopathy-M protein-skin lesions (POEMS) syndrome, and subjects with myeloma and amyloidosis will be eligible if they have measurable disease as defined above.
5. Subjects must have completed their most recent drug therapy directed at multiple myeloma in the following timeframes: * Chemotherapy, biological therapy, immunotherapy, or an investigational therapy at least 2 weeks prior to starting DS3032b; * Corticosteroids at least 2 weeks prior to starting DS3032b, except for a dose equivalent to dexamethasone of >/=4 mg/day; * Nitrosoureas, nitrogen mustards, mitomycin C, or monoclonal antibodies at least 6 weeks prior to starting DS3032b; * Autologous stem cell transplantation at least 12 weeks prior to starting DS3032b; * Allogeneic stem cell transplantation at least 24 weeks prior to starting DS3032b, and these subjects must also NOT have moderate to severe active acute or chronic graft versus host disease (GVHD).
6. #5 cont...* Previous and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted if such therapy has not been changed within 8 weeks before study drug treatment.
7. Subjects >/= 18 years old
8. Subjects must have Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
9. Subjects must have evidence of adequate hepatic function, as defined by the following: aspartate aminotransferase (AST)/alanine transaminase (ALT) <3 x upper limit of normal (ULN); Bilirubin </=1.5 xULN unless known to have Gilbert's syndrome or elevated bilirubin resulting from hemolysis
10. Subjects must have evidence of adequate bone marrow reserves, as defined by the following: Absolute neutrophil count (ANC) >/=1,000 cells/mm^3 without growth factors within 1 week of the initiation of treatment; Hemoglobin >/=8 g/dL without red blood cell transfusions within 2 weeks of the initiation of treatment; Platelet count >/=70,000 cells/mm^3 if marrow plasmacytosis < 50%. Platelet count >/=30,000 cells/mm^3 if marrow plasmacytosis >/= 50%.
11. 10. Subjects must have evidence of adequate renal function, as defined by the following: Serum creatinine within the institutional normal limits, OR if the creatinine is elevated: Creatinine clearance (CrCl) >/=30 mL/min., as measured by a 24-hour urine collection, or estimated by the Cockcroft and Gault formula: i. Female CrCl=[(140 - age in years) x weight in kg x 0.85]/(72 x serum creatinine in mg/dL) ii. Male CrCl = [(140 - age in years) x weight in kg x 1.00]/(72 x serum creatinine in mg/dL)
12. Subjects must have adequate blood clotting function, defined as International normalized ratio (INR) and activated partial thromboplastin time (aPTT) </= 1.5 x ULN
13. Subjects must have evidence of adequate cardiac function, as defined by the following: Absence of New York Heart Association (NYHA) class II, III, or IV congestive heart failure Absence of uncontrolled angina or hypertension; Absence of myocardial infarction in the previous 6 months; Absence of clinically significant bradycardia, or other uncontrolled cardiac arrhythmia defined as grade 3 or 4 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
14. Subjects who have received radiation therapy targeting > 10% of the bone marrow space must have completed this at least 2 weeks prior to starting therapy with DS3032b.
15. Subjects who have undergone any recent major surgery must have done so at least 4 weeks prior to starting therapy with DS3032b, with the following exceptions: Vertebroplasty and/or kyphoplasty, which must have been performed at least 1 week prior to starting DS3032b; Planned elective surgery unrelated to the subject's diagnosis of multiple myeloma, such as hernia repair, may be allowed, at the discretion of the Principle Investigator, as long as it was performed at least 2 weeks prior to starting DS3032b, and subjects have recovered fully from this procedure
16. Subject must be able to provide written informed consent, comply with protocol visits and procedures, and take oral medication, and does not have any active infection or comorbidity that would interfere with therapy.
17. Subjects (male and female) of childbearing/reproductive potential must agree to use double barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug.
18. Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects).
19. Subjects must sign and date an Institutional Review Board-approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study-specific procedures or tests.
20. Subjects must be able and willing to provide bone marrow biopsies/aspirates as requested by the protocol.
21. Subjects must be willing to undergo malignancy genotyping for TP53 mutation, insertion, or deletion at screening.
22. Subjects must have an estimated life expectancy of at least 3 months.

Exclusion Criteria:

1. Subjects who are receiving any concurrent investigational or conventional agent with known or suspected activity against multiple myeloma, or those whose adverse events due to agents administered more than 4 weeks earlier have not recovered to a severity of grade 0 or grade 1. Subjects with chronic Grade 2 toxicities may be eligible per discretion of the Investigator and MDACC investigational new drug (IND) Office (eg, Grade 2 chemotherapy-induced neuropathy).
2. Subject who received any therapies intended to treat malignancy within 21 days of first receipt of DS-3032b
3. Subjects with a malignancy that contains a non-synonymous mutation, insertion, or deletion in the TP53 gene determined previously or at screening.
4. Subjects with known central nervous system involvement with multiple myeloma will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. Subjects with a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to DS3032b.
6. Subjects with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, in the opinion of the Principal Investigator.
7. Subjects who are pregnant or breast-feeding
8. Subjects with an uncontrolled infection requiring intravenous antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or active hepatitis A, B or C infection.
9. Subjects with gastrointestinal conditions that could affect the absorption of DS-3032b in the opinion of the Investigator.
10. Subjects with prolongation of corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is >450 milliseconds (ms) for males and > 470 ms for females based on electrocardiogram (ECG).
11. Subjects who have required plasmapheresis and exchange less than 2 weeks prior to initiation of therapy with DS3032b.
12. Subjects with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Subjects are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years, and are considered by their physician to be at less than 30% risk of relapse. In addition, subjects with basal or squamous cell carcinoma of the skin, superficial carcinoma of the bladder, carcinoma of the prostate with a current prostate-specific antigen (PSA) value of <0.5 ng/mL, or cervical intraepithelial neoplasia will be eligible. Finally, subjects who are on hormonal therapy for a history of either prostate cancer or breast cancer may enroll, provided that there has been no evidence of disease progression during the previous three years.
13. Substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
14. Subjects with prior treatment with an MDM2 inhibitor.
15. Nonclinical studies indicate that DS-3032b is metabolized by CYP3A4/5. Drugs that are strong inhibitors or inducers of these enzymes may alter the PK of DS-3032b and should therefore be avoided. St. John's wort (hypericin) therefore will not be permitted for 30 days before and during participation in the study. Because DS-3032b is a substrate for CYP3A4/5 and grapefruit juice is a CYP3A4/5 inhibitor, foods or beverages containing grapefruit should not be taken within 48 hours before initial dose of study drug and throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of DS-3032b in Participants with Relapsed and/or Refractory Myeloma | 28 days
  MTD defined as the highest dose at which six subjects have been treated and less than two subjects experienced dose limiting toxicity (DLT) within the first cycle of treatment. DLT defined as any treatment-emergent adverse event (TEAE) not attributable to disease or disease-related processes that occurs during the observation period (Cycle 1) in each dose-level cohort per NCI-CTCAE v4.

SECONDARY OUTCOMES:
Response of DS-3032b in Participants with Relapsed and/or Refractory Myeloma | Every 28 days while participant is on the study
  Response determined by the IMWG Uniform Response Criteria and updated uniform response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hans C. Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org